CLINICAL TRIAL: NCT02350413
Title: Multicenter Italian Validation of EHP-30 at Centres Located in the Territory
Brief Title: Multicenter Italian Validation of EHP-30
Status: Completed | Type: Observational
Sponsor: University of Cagliari (Other)
Collaborators: University of Siena (Other); University of Foggia (Other); University of Padova (Other); University of Pisa (Other); Santa Chiara Hospital (Other)
Responsible Party: Principal Investigator, Stefano Angioni, Associate Professor, University of Cagliari
Other Study IDs: ENDOCA1415
Record Dates: First submitted 2015-01-13; First posted 2015-01-29 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Endometriosis; Quality of Life
MeSH Terms: conditions — Endometriosis | interventions — 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Endometriosis: Women referred to five Obstetrics and Gynecological Department for the treatment of endometriosis
  Interventions: Other: The Endometriosis Health Profile EPH-30

INTERVENTIONS:
Other: The Endometriosis Health Profile EPH-30 — Self-reported questionnaires
  Other Names: Sf 36; HADS; BAT; FSFI; Biberglou's scale; VAS Pain

SUMMARY:
The experience of the chronic illness negatively engraves on the quality of life of patients. Endometriosis is a disease that affects millions of women of childbearing age; it has repercussions on psychological health, as shown by numerous recent studies.

The aim of the present study is to validate the italian version of EPH 30, a self reported questionnaire, already used internationally, in order to determine the quality of life in women with endometriosis, assess their psychological health and the effectiveness of therapies.

ELIGIBILITY:
Inclusion Criteria:

* Previous surgical and histological diagnosis of endometriosis

Exclusion Criteria:

* Severe underlying comorbidities (gynecological, cardiovascular, respiratory, renal, hematological, endocrine, hepatic, gastrointestinal, neurological)
* Psychiatric diseases
* Refusal or inability to sign the informed consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women referred to five Obstetrics and Gynecological Department for the treatment of endometriosis.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
EHP- 30 The Endometriosis Health Profile | Cases were administered and fulfilled the questionnaires at the moment of diagnosis of endometriosis up to 4 weeks
  The EHP is the only condition-specific PRO designed from the patient's perspective to assess health related quality of life in endometriosis.The core questionnaire is composed of 30 items grouped into five scales: pain (11 items), control & powerlessness (6 items), emotional well-being (6 items), social support (4 items), and self-image (3 items). The modular questionnaire is composed of 23 items grouped into 6 scales: work life (5 items), relationship with children (2 items), sexual inter- course (5 items), medical profession (4 items), treatment (3 items), and infertility (4 items). The modular question- naire is characterized by the possibility of responding only to scales which the patient deems relevant to her. All scales can achieve a minimum score of 0, indicating low disabil- ity, and a maximum score of 100, indicating high disabil- ity. All items of a scale must be answered to be able to calculate a scale score.
SF-36 BPS Short Form 36 Bodily Pain Scale | Cases were administered and fulfilled the questionnaires at the moment of diagnosis of endometriosis up to 4 weeks
  The SF-36 BPS assesses bodily pain intensity and interference of pain with normal activities The SF-36 BPS is a 2-item scale.Responses for each of the 2 SF-36 BPS items are recoded into final item values . The raw scale score is computed as a simple algebraic sum of the recoded item values. The raw scale score is then transformed to a 0-100 scale. Norm-based scores may be calculated for SF-36v2 by including population normative data in the scoring algorithms. The BPS score is only calculated if both items are completed.
  Score interpretation. SF-36v1 BPS scores range from 0-100. A higher score indicates lack of bodily pain. SF-36v2 uses norm-based scoring, where 50 is the "average" for the population. Therefore, scores above or below 50 can be considered above or below, respectively, the population average health status for bodily pain, and scores can be interpreted based on deviance from the mean (10 points = 1 SD). Population normative data are available for the US and UK
HADS Hospital Anxiety and Depression Scale | Cases were administered and fulfilled the questionnaires at the moment of diagnosis of endometriosis up to 4 weeks
  It is commonly used by doctors to determine the levels of anxiety and depression that a person is experiencing. The HADS is a fourteen item scale that generates ordinal data. Seven of the items relate to anxiety and seven relate to depression.This, it was hoped, would create a tool for the detection of anxiety and depression in people with physical health problems.Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. The HADS uses a scale and therefore the data returned from the HADS is ordinal. Do Higher scores represent a worse outcome and is noted that the patient suffers from depression and anxiety
BAT Body Attitude Test | Cases were administered and fulfilled the questionnaires at the moment of diagnosis of endometriosis up to 4 weeks
  is a self-report questionnaire composed of 20 items and is aimed at measuring the participant's attitude toward their body, while effectively detecting cases of negative body perception even when not associated with eating disorders. This ques- tionnaire is thought to measure three areas of body experience mainly: (a) negative apprecia- tion of body size (Fact 1); (b) lack of familiarity with one's own body (Fact 2); and (c) general body dissatisfaction (Fact 3). High scores (maxi- mum is 100) correspond to a higher degree of body dissatisfaction
FSFI Female Sexual Function Index | Cases were administered and fulfilled the questionnaires at the moment of diagnosis of endometriosis up to 4 weeks
  self-reporting questionnaire made up of 19 items evaluating six domains: desire, arousal, lubrication, orgasm, satisfaction, and pain. The full-scale score is a minimum of 2.0 and a maximum of 36.0 and is obtained by adding the scores of each of the domains. A low score is significant for decreased sexual function, but for the pain domain, low scores indicate greater pain.
VAS PAIN Visual Analog Scale for Pain | Cases were administered and fulfilled the questionnaires at the moment of diagnosis of endometriosis up to 4 weeks
  The pain VAS is a continuous scale comprised of a horizontal (HVAS) or vertical (VVAS) line, usually 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme.For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale])A higher score indicates greater pain intensity. Based on the distribution of pain VAS scores in postsurgical patients ( hysterectomy, or laparoscopic myomectomy) who described their postoperative pain intensity as none, mild, moderate, or severe, the following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75- 100 mm)
Biberoglu and Behrman scale | Cases were administered and fulfilled the questionnaires at the moment of diagnosis of endometriosis up to 4 weeks
  The Biberoglu and Behrman scale consists of three patient-reported symptoms (dysmenorrhea, dyspareunia, and pelvic pain not related to menses) and two signs assessed during pelvic examination (pelvic tenderness and induration). Each of which are graded on a scale from 0 to 3 (or 4), with higher numbers indicating more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Angioni, MD, PhD, Principal Investigator — University of Cagliari
Locations (1):
- University of Cagliari,Obstetrics and Gynecological Department,, Monserrato, Cagliari, Italy